CLINICAL TRIAL: NCT02294864
Title: A Controlled Comparison of Pulsed Radiofrequency Vs Physical Therapy on Treating Chronic Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Long Beach Healthcare System (U.S. Federal Agency)
Collaborators: Southern California Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Ravi Mirpuri, University Of California Resident Physician, VA Long Beach Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #1283
Record Dates: First submitted 2014-11-12; First posted 2014-11-19 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Knee Osteoarthritis
Keywords: focus: pulsed radiofrequency (E02.779.468.599)
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Pulsed Radiofrequency Treatment; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulsed Radiofrequency (Experimental): Pulsed Radiofrequency This group will receive one dose of intra-articular PRF in the affected knee using previous literature standards. This includes standard blood pressure monitoring, sterile preparation, and needle insertion of the PRF probe directed at the site of maximal pain. The RFG-3C Plus radiofrequency generator will be activated at 42C, pulse width 10ms, and 2Hz frequency for 15 min.
  Interventions: Device: Percutaneous Pulsed Radiofrequency
- Physical Therapy (Active Comparator): This group will receive standard of care outpatient physical therapy weekly for 3-4 weeks with therapist instructions to reduce knee pain.
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Device: Percutaneous Pulsed Radiofrequency — Pulsed Radiofrequency
  Other Names: Pulsed Radiofrequency
  Arms: Pulsed Radiofrequency
Procedure: Physical Therapy
  Other Names: Physical Therapy for 4 weeks
  Arms: Physical Therapy

SUMMARY:
It is estimated that nearly 27 million US adults have osteoarthritis (OA) and suffer from pain . Pulsed Radio Frequency (PRF) is one method that has been successfully used in treatment of various etiologies of pain. However there are limited studies and research that prove its effectiveness in treating articular pain. The proposed study's primary aim is determining if PRF is an effective treatment for chronic osteoarthritic knee pain. This study hypothesizes that PRF has analgesic properties immediately after treatment and at least 3 months afterwards compared to control treatment with physical therapy.

Additionally this research project addresses several other objectives including:

1. Provide a controlled study to determine the effectiveness of PRF for intra-articular pain
2. Determine how effective PRF is 1 month and 3 months after treatment for articular pain.
3. Further scientific evidence on the overall effectiveness of PRF
4. Provide evidence that PRF likely has other mechanism of action besides direct nerve stimulation of inhibitory pain pathways.
5. Compare the effectiveness of PRF vs Physical Therapy in treating chronic knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18
* Radiologic evidence of Kellgren-Lawrence knee arthritis between levels 1-3
* Satisfy the American College of Rheumatology criteria for knee osteoarthritis.

Exclusion Criteria:

* Failure to satisfy inclusion criteria
* Existence of general contraindications against percutaneous knee intervention including (e.g. infection, hemorrhagic diathesis, anticoagulated patients)
* Patients with pacemaker or stimulator implants
* Metallic hardware located in the treatment knee of choice
* High clinical suspicion for alternative diagnosis other than Knee Osteoarthritis
* VA defined vulnerable populations (e.g. adults with cognitive impairments, mentally retarded, non-english speaking, severe psychiatric disorders, prisoners, terminally ill patient, employees, homeless, pregnant).
* Any patient that would not be able to follow up at 1 and 3 months after intervention.
* Any patient unwilling to receive physical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
VAS pain scores and Western Ontario and McMaster Universities Arthritis Index (WOMAC) with pulsed radiofrequency vs physical therapy | 3 months
  The Study will measure VAS pain scores (0-10) at initial consult, 1 month, and 3 months. Additionally the study will document functional changes using the WOMAC questionnaire at initial evaluation and 3 months.

SECONDARY OUTCOMES:
Safety of pulsed radiofrequency for knee pain treatment | 3 months
  The study will measure and document any adverse effects that occur in the study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Takemoto, M.D., Principal Investigator — Principal Investigator; Ravi Mirpuri, D.O., Principal Investigator — Long Beach VA resident
Locations (1):
- Long Beach Veterans Hospital, Long Beach, California, United States

REFERENCES:
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Guo L, Kubat NJ, Nelson TR, Isenberg RA. Meta-analysis of clinical efficacy of pulsed radio frequency energy treatment. Ann Surg. 2012 Mar;255(3):457-67. doi: 10.1097/SLA.0b013e3182447b5d. PMID 22301609
- [Background] Sluijter ME, Teixeira A, Serra V, Balogh S, Schianchi P. Intra-articular application of pulsed radiofrequency for arthrogenic pain--report of six cases. Pain Pract. 2008 Jan-Feb;8(1):57-61. doi: 10.1111/j.1533-2500.2007.00172.x. No abstract available. PMID 18211593
- [Background] Karaman H, Tufek A, Kavak GO, Yildirim ZB, Uysal E, Celik F, Kaya S. Intra-articularly applied pulsed radiofrequency can reduce chronic knee pain in patients with osteoarthritis. J Chin Med Assoc. 2011 Aug;74(8):336-40. doi: 10.1016/j.jcma.2011.06.004. Epub 2011 Jul 23. PMID 21872812